CLINICAL TRIAL: NCT00969709
Title: A Double-blind, Placebo-Controlled, Fixed-Dose Study of F2695 SR in Patients With Major Depressive Disorder
Brief Title: Safety and Efficacy of Levomilnacipran ER (F2695 SR) in Major Depressive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LVM-MD-01
Record Dates: First submitted 2009-08-31; First posted 2009-09-01 (Estimated); Results first posted 2013-10-25 (Estimated); Last update posted 2013-10-25 (Estimated); Status verified 2013-08

CONDITIONS: Major Depressive Disorder
Keywords: Depression; Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Levomilnacipran

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): 40 mg Levomilnacipran ER capsules, low dose, oral administration, once daily.
  Interventions: Drug: Levomilnacipran ER
- 2 (Experimental): 80 mg Levomilnacipran ER capsules, medium dose, oral administration, once daily dosing
  Interventions: Drug: Levomilnacipran ER
- 3 (Experimental): 120 mg Levomilnacipran ER capsules, high dose, oral administration, once daily dosing
  Interventions: Drug: Levomilnacipran ER
- 4 (Placebo Comparator): Matching placebo capsules, oral administration, once daily.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Levomilnacipran ER — Levomilnacipran ER, 40 mg, oral administration, in capsule form, once daily for 8 weeks.
  Arms: 1
Drug: Levomilnacipran ER — Levomilnacipran ER, 80 mg, oral administration, in capsule form, once daily for 8 weeks.
  Arms: 2
Drug: Levomilnacipran ER — Levomilnacipran ER, 120 mg, oral administration, in capsule form, once daily for 8 weeks.
  Arms: 3
Drug: Placebo — Matching placebo capsules, oral administration, once daily for 8 weeks.
  Arms: 4

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety, and tolerability of Levomilnacipran ER fixed doses versus placebo in the treatment of outpatients with major depressive disorder.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, 18-65 years old
* Currently meet the DSM-IV-TR criteria for Major Depressive Disorder
* The patient's current depressive episode must be at least 8 weeks in duration

Exclusion Criteria:

* Women who are pregnant, women who will be breastfeeding during the study, and women with childbearing potential who are not practicing a reliable method of birth control
* Patients with a history of meeting DSM-IV-TR criteria for:

  * any manic or hypomanic episode
  * schizophrenia or any other psychotic disorder
  * obsessive-compulsive disorder
* Patients who are considered a suicide risk

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 724 (Actual)
Dates: Start 2009-09; Primary Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carl Gommoll, MS, Study Director — Forest Research Institute, a subsidiary of Forest Laboratories Inc.
Locations (36):
- United States (36):
  - Forest Investigative Site, Phoenix, Arizona
  - Forest Investigative Site, Scottsdale, Arizona
  - Forest Investigative Site, Beverly Hills, California
  - Forest Investigative Site, Costa Mesa, California
  - Forest Investigative Site, Escondido, California
  - Forest Investigative Site, Oceanside, California
  - Forest Investigative Site, Sherman Oaks, California
  - Forest Investigative Site, Denver, Colorado
  - Forest Investigative Site, Cromwell, Connecticut
  - Forest Investigative Site, Coral Springs, Florida
  - Forest Investigative Site, Fort Myers, Florida
  - Forest Investigative Site, Hallandale, Florida
  - Forest Investigative Site, Jacksonville, Florida
  - Forest Investigative Site, Orlando, Florida
  - Forest Investigative Site, West Palm Beach, Florida
  - Forest Investigative Site, Hoffman Estates, Illinois
  - Forest Investigative Site, Wichita, Kansas
  - Forest Investigative Site, Baltimore, Maryland
  - Forest Investigative Site, Rockville, Maryland
  - Forest Investigative Site, Cherry Hill, New Jersey
  - Forest Investigative Site, Willingboro, New Jersey
  - Forest Investigative Site, Brooklyn, New York
  - Forest Investigative Site, Mount Kisco, New York
  - Forest Investigative Site, New York, New York
  - Forest Investigative Site, Staten Island, New York
  - Forest Investigative Site, Raleigh, North Carolina
  - Forest Investigative Site, Canton, Ohio
  - Forest Investigative Site, Portland, Oregon
  - Forest Investigative Site, Media, Pennsylvania
  - Forest Investigative Site, Norristown, Pennsylvania
  - Forest Investigative Site, Lincoln, Rhode Island
  - Forest Investigative Site, Memphis, Tennessee
  - Forest Investigative Site, Dallas, Texas
  - Forest Investigative Site, San Antonio, Texas
  - Forest Investigative Site, Bellevue, Washington
  - Forest Investigative Site, Seattle, Washington

REFERENCES:
- [Derived] Cutler AJ, Gommoll CP, Chen C, Greenberg WM, Ruth A. Levomilnacipran Extended-Release Treatment in Patients With Major Depressive Disorder: Improvements in Functional Impairment Categories. Prim Care Companion CNS Disord. 2015 Jun 11;17(3):10.4088/PCC.14m01753. doi: 10.4088/PCC.14m01753. eCollection 2015. PMID 26644957
- [Derived] Blum SI, Tourkodimitris S, Ruth A. Evaluation of functional health and well-being in patients receiving levomilnacipran ER for the treatment of major depressive disorder. J Affect Disord. 2015 Jan 1;170:230-6. doi: 10.1016/j.jad.2014.09.005. Epub 2014 Sep 10. PMID 25259674
- [Derived] Asnis GM, Bose A, Gommoll CP, Chen C, Greenberg WM. Efficacy and safety of levomilnacipran sustained release 40 mg, 80 mg, or 120 mg in major depressive disorder: a phase 3, randomized, double-blind, placebo-controlled study. J Clin Psychiatry. 2013 Mar;74(3):242-8. doi: 10.4088/JCP.12m08197. PMID 23561229

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient recruitment at 38 study centers located in the United States during a 17 month period from September 2009 to February 2011.
Pre-assignment Details: The study included a 1-week, single-blind placebo run-in period immediately before the 8-week double-blind treatment period.
Groups:
- Placebo: Dose matching placebo capsules, oral administration, once daily dosing.
  Placebo : Matching placebo capsules, oral administration, once daily for 8 weeks.
- Levomilnacipran ER 40 mg: 40 mg/day Levomilnacipran ER capsules, low dose, oral administration, once daily dosing.
  Levomilnacipran ER, low dose, oral administration, in capsule form, once daily for 8 weeks.
- Levomilnacipran ER 80 mg: 80 mg/day Levomilnacipran ER capsules, medium dose, oral administration, once daily dosing
  Levomilnacipran ER, medium dose, oral administration, in capsule form, once daily for 8 weeks.
- Levomilnacipran ER 120 mg: 120 mg/day Levomilnacipran ER capsules, high dose, oral administration, once daily dosing
  Levomilnacipran ER, high dose, oral administration, in capsule form, once daily for 8 weeks.
Period: Overall Study
Arm/Group | Placebo | Levomilnacipran ER 40 mg | Levomilnacipran ER 80 mg | Levomilnacipran ER 120 mg
Started | 176 | 178 | 179 | 180
Completed | 138 | 130 | 121 | 117
Not Completed | 38 | 48 | 58 | 63
Not completed — Adverse Event | 3 | 13 | 26 | 12
Not completed — Lack of Efficacy | 7 | 4 | 1 | 3
Not completed — Protocol Violation | 9 | 5 | 9 | 10
Not completed — Withdrawal by Subject | 9 | 12 | 11 | 23
Not completed — Lost to Follow-up | 10 | 14 | 8 | 15
Not completed — Other reasons | 0 | 0 | 3 | 0

BASELINE CHARACTERISTICS:
Population: A total of 724 patients were randomized to receive double-blind treatment (Randomized Population); 713 patients received at least 1 dose of treatment (Safety Population). The demographic analyses of the baseline participants is based on the Safety Population
Groups:
- Placebo: Dose matching placebo capsules, oral administration, once daily dosing for 8 weeks
- Levomilnacipran ER 40 mg: 40 mg per day Levomilnacipran ER capsules, oral administration, once daily for 8 weeks.
- Levomilnacipran ER 80 mg: 80 mg per day Levomilnacipran ER capsules, oral administration, once daily for 8 weeks.
- Levomilnacipran ER 120 mg: 120 mg per day Levomilnacipran ER capsules, oral administration, once daily for 8 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | Levomilnacipran ER 40 mg | Levomilnacipran ER 80 mg | Levomilnacipran ER 120 mg | Total
Number analyzed (Participants) | 176 | 178 | 179 | 180 | 713
Age Continuous [Mean (Standard Deviation); unit: years] | 43.1 (11.3) | 41.6 (13.1) | 41.0 (12.8) | 40.3 (11.9) | 41.1 (12.3)
Age, Customized [Number; unit: participants]
  18 years to 19 years | 1 | 2 | 4 | 2 | 9
  20 years to 29 years | 31 | 43 | 44 | 42 | 160
  30 years to 39 years | 47 | 34 | 33 | 38 | 152
  40 years to 49 years | 44 | 36 | 48 | 46 | 174
  50 years to 59 years | 46 | 48 | 36 | 41 | 171
  60 years to 65 years | 7 | 15 | 14 | 11 | 47
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 108 | 122 | 111 | 106 | 447
  Male | 68 | 56 | 68 | 74 | 266
Race/Ethnicity, Customized [Number; unit: participants]
  White | 134 | 133 | 129 | 130 | 526
  Black or African American | 29 | 36 | 39 | 41 | 145
  Asian | 8 | 3 | 5 | 3 | 19
  American Indian or Alaska native | 1 | 0 | 2 | 1 | 4
  Native Hawaiian or other Pacific Islander | 0 | 0 | 0 | 1 | 1
  Other | 3 | 6 | 4 | 4 | 17
  Hispanic or Latino | 20 | 22 | 28 | 22 | 92
  Not Hispanic or Latino | 156 | 155 | 151 | 158 | 620
Region of Enrollment [Number; unit: participants]
  United States | 176 | 178 | 179 | 180 | 713
Weight [Mean (Standard Deviation); unit: kg] | 83.8 (19.3) | 79.5 (17.1) | 83.0 (17.3) | 84.2 (18.6) | 82.6 (18.1)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: Kilograms Per Meter Squared] | 29.0 (5.8) | 28.0 (5.3) | 28.9 (5.4) | 29.2 (5.4) | 28.8 (5.5)

OUTCOME MEASURES:

1. Primary Outcome: Change in Montgomery-Åsberg Depression Rating Scale (MADRS) Total Score
Description: The MADRS was used to assess depressive symptomatology during the past week. Patients are rated on 10 items to assess feelings of sadness, lassitude, pessimism, inner tension, suicidality, reduced sleep or appetite, difficulty concentrating, and lack of interest.
  Each item of the 10 items are scored on a 7-point scale. A score of 0 indicates the absence of symptoms,and a score of 6 indicates symptoms of maximum severity. The total MADRS score for this measure ranges from 0 (absence of symptoms) to 60 (maximum severity for all measured symptoms).
Time Frame: From Baseline to Week 8
Population: A total of 724 patients were randomized to receive double-blind treatment (Randomized Population); 713 patients received at least 1 dose of treatment (Safety Population); and 704 patients received at least 1 dose of treatment and had at least 1 postbaseline MADRS-CR assessment (Intent to Treat [ITT] Population).
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Levomilnacipran ER 40 mg | Levomilnacipran ER 80 mg | Levomilnacipran ER 120 mg
Number analyzed (Participants) | 175 | 176 | 177 | 176
Units on a scale | -11.6 (0.97) | -14.8 (0.99) | -15.6 (1.00) | -16.5 (1.02)
Statistical Analysis 1: Comparison: Placebo vs Levomilnacipran ER 40 mg; Test type: Superiority or Other; p = 0.0186, Mixed Models Analysis; Mixed-effects model for repeated measures; Least squares mean difference = -3.23, 95% CI 2-sided [-5.92 to -0.54]
Statistical Analysis 2: Comparison: Placebo vs Levomilnacipran ER 80 mg; Test type: Superiority or Other; p = 0.0038, Mixed Models Analysis; Mixed-effects model for repeated measures; Least squares mean difference = -3.99, 95% CI 2-sided [-6.69 to -1.29]
Statistical Analysis 3: Comparison: Placebo vs Levomilnacipran ER 120 mg; Test type: Superiority or Other; p = 0.0005, Mixed Models Analysis; Mixed-effects model for repeated measures; Least squares mean difference = -4.86, 95% CI 2-sided [-7.59 to -2.12]

2. Secondary Outcome: Change in Sheehan Disability Scale (SDS) Total Score
Description: The Sheehan Disability Scale (SDS) is a 3-item clinician-rated questionnaire used to evaluate functional impairments in the domains of work, social life/leisure, and family life/home responsibility. All items are rated on an 11-point continuum (0 = no impairment to 10 = most severe) with the total SDS score ranging from 0 (no impairment) to 30 (most severe for all measured symptoms)
Time Frame: From Baseline to Week 8
Population: A total of 724 patients were randomized to receive double-blind treatment (Randomized Population); 713 patients received at least 1 dose of treatment (Safety Population); and 704 patients received at least 1 dose of treatment and had at least 1 postbaseline MADRS-CR assessment(Intent to Treat [ITT] Population).
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Levomilnacipran ER 40 mg | Levomilnacipran ER 80 mg | Levomilnacipran ER 120 mg
Number analyzed (Participants) | 175 | 176 | 177 | 176
units on a scale | -7.2 (0.74) | -8.6 (0.75) | -9.7 (0.77) | -9.7 (0.78)
Statistical Analysis 1: Comparison: Placebo vs Levomilnacipran ER 40 mg; Test type: Superiority or Other; p = 0.1687, Mixed Models Analysis; Mixed-effects model for repeated measures; Least squares mean difference = -1.41, 95% CI 2-sided [-3.42 to 0.60]
Statistical Analysis 2: Comparison: Placebo vs Levomilnacipran ER 80 mg; Test type: Superiority or Other; p = 0.0151, Mixed Models Analysis; Mixed-effects model for repeated measures; least squares mean difference = -2.51, 95% CI 2-sided [-4.54 to -0.49]
Statistical Analysis 3: Comparison: Placebo vs Levomilnacipran ER 120 mg; Test type: Superiority or Other; p = 0.0141, Mixed Models Analysis; Mixed-effects model for repeated measures; Least squares mean difference = -2.57, 95% CI 2-sided [-4.62 to -0.52]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over a 20 month period from September 2009 to June 2011 at 38 study sites.
Description: The Serious Adverse Event data presented here is for the safety population. The Other Adverse Event data presented here is for the safety population during the 8 week double-blind treatment period.
Groups:
- Levomilnacipran ER 40 mg: 40 mg per day Levomilnacipran ER, low dose, oral administration, once daily for 8 weeks.
Arm/Group | Placebo | Levomilnacipran ER 40 mg | Levomilnacipran ER 80 mg | Levomilnacipran ER 120 mg
Serious Adverse Events (participants affected / at risk) | 1/176 | 3/178 | 2/179 | 1/180
Other Adverse Events (participants affected / at risk) | 66/176 | 110/178 | 122/179 | 112/180
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Placebo (N=176) | Levomilnacipran ER 40 mg (N=178) | Levomilnacipran ER 80 mg (N=179) | Levomilnacipran ER 120 mg (N=180)
Aggression (Psychiatric disorders) | 0 | 1 | 0 | 0
Chest Pain (General disorders) | 0 | 1 | 0 | 0
Cytomegalovirus mononucleosis (Infections and infestations) | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Suicide Attempt (Psychiatric disorders) | 0 | 1 | 0 | 0
Premature baby (Pregnancy, puerperium and perinatal conditions) | 0/108 | 0/122 | 0/111 | 1/106
Small for dates baby (Pregnancy, puerperium and perinatal conditions) | 0/108 | 0/122 | 0/111 | 1/106
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 0/108 | 0/122 | 1/111 | 0/106
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Placebo (N=176) | Levomilnacipran ER 40 mg (N=178) | Levomilnacipran ER 80 mg (N=179) | Levomilnacipran ER 120 mg (N=180)
Headache (Nervous system disorders) | 20 | 29 | 36 | 27
Nausea (Gastrointestinal disorders) | 4 | 19 | 39 | 23
Constipation (Gastrointestinal disorders) | 7 | 19 | 18 | 23
Dry mouth (Gastrointestinal disorders) | 17 | 20 | 12 | 27
Heart rate increased (Investigations) | 3 | 18 | 11 | 17
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 | 9 | 24 | 10
Dizziness (Nervous system disorders) | 8 | 10 | 17 | 14
Upper respiratory tract infection (Infections and infestations) | 10 | 14 | 11 | 4
Nasopharyngitis (Infections and infestations) | 10 | 11 | 9 | 7
Palpitations (Cardiac disorders) | 1 | 8 | 11 | 8
Vomiting (Gastrointestinal disorders) | 0 | 10 | 10 | 6
Insomnia (Psychiatric disorders) | 7 | 7 | 11 | 7
Urinary hesitation (Renal and urinary disorders) | 0 | 7 | 6 | 11
Diarrhoea (Gastrointestinal disorders) | 3 | 8 | 7 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 2 | 9 | 7
Tachycardia (Cardiac disorders) | 0 | 4 | 11 | 3
Erectile dysfunction (Reproductive system and breast disorders) | 2/68 | 3/56 | 2/68 | 7/74
Ejaculation delayed (Reproductive system and breast disorders) | 0/68 | 0/56 | 4/68 | 0/74

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All data generated in this study will be the property of Forest Research Institute, Inc. An integrated clinical and statistical report will be prepared at the completion of the study.

Publication of the results by the Investigator will be subject to mutual agreement between the Investigator and Forest Research Institute, Inc.